CLINICAL TRIAL: NCT00994084
Title: Healthy Kids-Houston: An Integrated Community Program for the Prevention of Obesity Among Minority Children
Brief Title: Healthy Kids-Houston: A Community Childhood Obesity Intervention Program
Acronym: HKH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, William Wong, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 26490-1; 2008-55215-18875
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Obesity
Keywords: Obesity; Minority children; Community intervention program; Lifestyle changes; Physical activities; Nutrition lessons; Behavior modification
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle modification (Active Comparator): This arm receives the intervention program that includes structured physical activities and nutrition and behavior lessons
  Interventions: Behavioral: Healthy Kids-Houston program
- Control (Placebo Comparator): This arm receives no intervention
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Healthy Kids-Houston program — Children receive 90 minutes of after-school structured physical activities and 30 minutes of nutrition and behavior lessons twice a week during three 6-week sessions at the community centers. The 6-week sessions take place once in the fall, once in early spring and once in late spring.
  Other Names: Healthy Kids-Houston curriculum
  Arms: Lifestyle modification
Behavioral: Control — Children do not receive the Healthy Kids-Houston behavior modification program but will participate in the regular after-school enrichment programs offered by the community centers.
  Arms: Control

SUMMARY:
The collaborative study is to determine the effectiveness of an after-school community-based program to prevent obesity among minority children.

DETAILED DESCRIPTION:
Childhood obesity is a major health issue in the United States, particularly among minority children. An integrated after-school program that offers structured and fun physical activities with nutrition and behavior lessons in community centers operated by the Houston Parks and Recreation Department might prevent obesity among minority children who live in the neighborhood.

ELIGIBILITY:
Inclusion Criteria:

* Live in close proximity of the community centers

Exclusion Criteria:

* Medical or physical conditions that prevent the child from participating in the physical activities

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1094 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Body mass index | One school year

SECONDARY OUTCOMES:
Agility | One school year
Muscular strength and endurance | One school year
Self esteem | One school year
Physical activity level | One school year
Flexibility | One school year

CONTACTS AND LOCATIONS:
Overall Officials: William W Wong, PhD, Study Director — Baylor College of Medicine
Locations (1):
- Houston Parks and Recreation Department Community Centers, Houston, Texas, United States

REFERENCES:
- [Background] Wong WW, Mikhail C, Ortiz CL, Lathan D, Moore LA, Konzelmann KL, Smith EO. Body weight has no impact on self-esteem of minority children living in inner city, low-income neighborhoods: a cross-sectional study. BMC Pediatr. 2014 Jan 24;14:19. doi: 10.1186/1471-2431-14-19. PMID 24456638
- [Result] Wong WW, Ortiz CL, Lathan D, Moore LA, Konzelmann KL, Adolph AL, Smith EO, Butte NF. Sleep duration of underserved minority children in a cross-sectional study. BMC Public Health. 2013 Jul 12;13:648. doi: 10.1186/1471-2458-13-648. PMID 23849231
- [Derived] Wong WW, Ortiz CL, Stuff JE, Mikhail C, Lathan D, Moore LA, Alejandro ME, Butte NF, Smith EO. A Community-based Healthy Living Promotion Program Improved Self-esteem Among Minority Children. J Pediatr Gastroenterol Nutr. 2016 Jul;63(1):106-12. doi: 10.1097/MPG.0000000000001088. PMID 27336592